CLINICAL TRIAL: NCT05100628
Title: A Dose Escalation and Dose Expansion Study of NOX66 Plus Doxorubicin in Anthracycline-naïve, Adult Patients With Soft Tissue Sarcoma - CEP-2
Brief Title: A Study of NOX66 Plus Doxorubicin in Anthracycline-naïve, Adult Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOX66-004
Record Dates: First submitted 2021-10-20; First posted 2021-10-29 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Soft-tissue Sarcoma
Keywords: Doxorubicin; Dose-escalation study; Dose-expansion study; Maximum tolerated dose
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin (Experimental)
  Interventions: Drug: NOX66; Drug: Doxorubicin
- Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin (Experimental)
  Interventions: Drug: NOX66; Drug: Doxorubicin
- Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin (Experimental)
  Interventions: Drug: NOX66; Drug: Doxorubicin
- Dose-Expansion Cohort: NOX66 + Doxorubicin (Experimental)
  Interventions: Drug: NOX66; Drug: Doxorubicin

INTERVENTIONS:
Drug: NOX66 — NOX66 800 mg (400 mg suppository twice daily [BID]).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Arms: Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin
Drug: NOX66 — NOX66 1200 mg daily (600 mg suppository BID).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Arms: Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin
Drug: NOX66 — NOX66 1800 mg daily (600 mg suppository thrice daily).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Arms: Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin
Drug: NOX66 — MTD of the combination of NOX66 and doxorubicin will be determined in the dose-escalation cohort of the study. The selected dose will be administered in combination with Doxorubicin.
  Arms: Dose-Expansion Cohort: NOX66 + Doxorubicin
Drug: Doxorubicin — Doxorubicin will be given at 75 mg/m^2 as an intravenous infusion on Day 2 of the 21-day cycle for up to 6 cycles.

SUMMARY:
This is a Phase I, open-label, dose-escalation and dose-expansion study of NOX66 given rectally, in cohorts of patients with metastatic soft tissue sarcoma (STS) who have not been exposed to anthracycline therapy, using a fixed dose-escalation schema every 21 days to establish the maximum tolerated dose (MTD) of the combination of NOX66 and doxorubicin.

DETAILED DESCRIPTION:
The study will contain dose-escalation cohorts and dose-expansion cohorts. The study design allows an exploration of different doses of NOX66 with safety monitoring to ensure the safety of the patients.

Dose-escalation cohorts: It will include three planned Treatment Groups (800, 1200, 1800 mg daily) and patients enrolled in these groups will receive 7 days of monotherapy treatment with NOX66 followed by a 5-day washout period. Thereafter, patients will enter a combination therapy (only if no significant toxicity is observed during monotherapy). This will commence with Cycle 1, which will consist of 7 days of NOX66, and on Day 2 of the 21-day cycle, doxorubicin will be administered. Patients will continue to be treated for up to 6 x 21-day cycles of NOX66 and doxorubicin. New patients will be entered at the next dose level of NOX66, if no dose-limiting toxicities have occurred among the first 3 patients at the end of cycle 1. During the dose-escalation, MTD of the combination of NOX66 and doxorubicin will be determined.

Dose-expansion cohort: On completion of the dose-escalation cohort, patients will be enrolled into a dose-expansion at the MTD of the combination of NOX66 and doxorubicin. All patients will enter directly into 21-day combination cycles and will be given NOX66 therapy for 7 days and doxorubicin will be administered on Day 2 of each cycle. Treatment will be terminated upon disease progression, unacceptable toxicity, or a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a histologically confirmed diagnosis of metastatic or recurrent soft tissue sarcoma
* Patients for whom treatment with doxorubicin is considered to be appropriate
* Left ventricular ejection fraction ≥ 50%
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Disease that is considered measurable according to RECIST v1.1.

Exclusion Criteria:

* Histologically or cytologically confirmed Kaposi's sarcoma, gastrointestinal stromal tumor (GIST), extra-skeletal myxoid chondrosarcoma, epithelioid hemangioendothelioma, and desmoid tumor
* Untreated metastases to the central nervous system
* Received previous treatment with anthracyclines and anthracenediones
* Previous radiation therapy to the mediastinal or pericardial area
* A known allergy to any of the treatment components
* Patient not willing to use suppositories
* Patients with a colostomy
* Patients who have had a colectomy (total or left hemicolectomy) with re-anastomosis
* Patients for whom administration of the suppositories are likely to cause pain (e.g., inflamed hemorrhoids, fissures, or lesions of the anus or rectum)
* Patients with fecal impaction, chronic idiopathic constipation, or chronic diarrhea or alternating irritable bowel disease
* Patients with inflammatory bowel disease
* Previous treatment with an investigational agent or the non-approved use of a drug or device within 4 weeks before study entry
* Uncontrolled diabetes mellitus
* Patients who require concomitant use of strong inhibitors or inducers of CYP3A4, CYP2D6 or P- glycoprotein (P- gp)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Mayo Clinic Florida - Oncology, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Site name Washington University School of Medicine in Saint Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were screened
Groups:
- Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin: NOX66: NOX66 800 mg (400 mg suppository twice daily [BID]).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Doxorubicin: Doxorubicin will be given at 75 mg/m^2 as an intravenous infusion on Day 2 of the 21-day cycle for up to 6 cycles.
- Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin: NOX66: NOX66 1200 mg daily (600 mg suppository BID).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Doxorubicin: Doxorubicin will be given at 75 mg/m^2 as an intravenous infusion on Day 2 of the 21-day cycle for up to 6 cycles.
- Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin: NOX66: NOX66 1800 mg daily (600 mg suppository thrice daily).
  Monotherapy: 7 days of NOX66 followed by 5 days washout. Combination therapy: 7 days of NOX66 followed by 14 days washout in a 21-day cycle, for up to 6 cycles.
  Doxorubicin: Doxorubicin will be given at 75 mg/m^2 as an intravenous infusion on Day 2 of the 21-day cycle for up to 6 cycles.
Period: Overall Study
Arm/Group | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin | Dose-Expansion Cohort: NOX66 + Doxorubicin
Started | 3 | 3 | 3 | 0
Completed | 2 | 2 | 0 | 0
Not Completed | 1 | 1 | 3 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 3 | 0
Not completed — unkown | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.07) | 52.0 (7.81) | 47.7 (17.57) | 51.3 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 0 | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 2 | 1 | 3 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Number of Patients With Dose-limiting Toxicities (DLTs)
Description: Determination of the MTD of NOX66 in combination with doxorubicin. MTD is defined as the dose level at which no more than 1 patient out of 6 experiences a DLT at the end of Cycle 1.
Time Frame: Cycle 1 of each dose (Cycle length is 21 days)
Population: Patients that received at least one dose of NOX66
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Adverse Events (AEs) for NOX66
Description: Characterization of the safety and tolerability of NOX66.
Time Frame: From first study treatment with DOX66 monotherapy through study completion, approximately of 14 months and 20 days. From February 11, 2022, to May 1, 2023
Population: Patients treated with at least one dose of NOX66
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  With at least one Adverse Event | 3 | 3 | 3
  With at least one TEAE (Treatment Emergent Adverse Event) | 3 | 3 | 3
  With at least one SAE | 1 | 1 | 0
  At least one TEAE possibly related to NOX66 | 3 | 2 | 1
  At least one TEAE related to NOX66 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All AEs and SAEs will be collected from the signing of the ICF until 30 days after the last dose of study drug, an average of 14 months.
Arm/Group | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin (N=3) | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin (N=3) | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation Cohort 1: NOX66 800 mg + Doxorubicin (N=3) | Dose-Escalation Cohort 2: NOX66 1200 mg + Doxorubicin (N=3) | Dose-Escalation Cohort 3: NOX66 1800 mg + Doxorubicin (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 2 (4) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (3) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT05100628/Prot_SAP_000.pdf